CLINICAL TRIAL: NCT01476449
Title: Monthly Ranibizumab Versus Treat and Extend Ranibizumab for Diabetic Macular Edema
Brief Title: Dosing Study of Ranibizumab for Diabetic Retinal and Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Retina Vitreous Associates of Florida (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1127228
Record Dates: First submitted 2011-11-13; First posted 2011-11-22 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Retinopathy; Macular Edema
Keywords: Diabetic Macular Edema; Diabetic Retinal Swelling; DIabetic Eye Disease
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monthly Ranibizumab (Active Comparator): Patients randomized to the Monthly Ranibizumab arm of the study will be administered intravitreal injections each month for their diabetic macular edema for the duration of the study.
  Interventions: Drug: Ranibizumab
- Treat and Extend Ranibizumab (Experimental): Patients randomized to this arm of the study will receive intravitreal injections of ranibizumab until their maculae are anatomically "dry," at which point the evaluation and injection interval will be extended.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Pars plana injection of ranibizumab 0.5mg into the vitreous cavity.
  Other Names: Lucentis
  Arms: Monthly Ranibizumab
Drug: Ranibizumab — Pars plana injection of ranibizumab 0.5mg into the vitreous cavity.
  Other Names: Lucentis
  Arms: Treat and Extend Ranibizumab

SUMMARY:
This study is to see whether treating diabetic retinal swelling with ranibizumab injections into the eye monthly is better than treating diabetic retinal swelling with ranibizumab injections into the eye less frequently.

DETAILED DESCRIPTION:
This is a prospective randomized study comparing two groups of patients with diabetic macular edema. One group will receive injections of ranibizumab monthly and the other group will have the option to receive injections of ranibizumab less frequently. That is eligible to receive the injections less frequently will have fewer injections given if the patients in that group are doing well.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Patient related considerations
* Phakic or pseudophakic patients with a known history of diabetes will be eligible.
* Women of reproductive age will be required to take a urine pregnancy test prior to administration of the study drug.
* Disease related considerations:
* Patients will have met standard, accepted diagnostic criteria for diabetes and will be currently treated with at least one systemic antihyperglycemic or insulin medication.
* Patients will have a BCVA ETDRS Snellen-equivalent less than or equal to 20/40
* Central foveal thickness on SD-OCT of >300um

Exclusion Criteria:

* Pregnancy (positive pregnancy test) or lactation Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Foveal ischemia on IVFA
* Intraocular surgery less than 6 months ago
* Epiretinal membrane of clinical significance
* Prior vitrectomy
* Uncontrolled glaucoma
* Macular or peripheral laser within 90 Days from Day 0 injection
* Intravitreal steroid injection within 90 days from Day 0 injection
* Intravitreal or systemic anti-VEGF within 30 days from Day 0 injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Eichenbaum, MD, Principal Investigator — Retina Vitreous Associates of Florida
Locations (2):
- United States (2):
  - Retina Vitreous Associates of Florida, Clearwater, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Monthly Ranibizumab | Treat and Extend Ranibizumab
Started | 10 | 10
Completed | 8 | 8
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monthly Ranibizumab | Treat and Extend Ranibizumab | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Full Range); unit: years] | 64.5 [53 to 86] | 60.4 [40 to 71] | 62.5 [40 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Early Treatment for Diabetic Retinopathy Study (ETDRS) Eye Chart Vision.
Description: The ETDRS eye chart was used to assess vision at each visit, with the change through month 24 reported.
Time Frame: Baseline through 24 months
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Monthly Ranibizumab | Treat and Extend Ranibizumab
Number analyzed (Participants) | 10 | 10
ETDRS Letters | 8.3 (7.2) | 8.5 (8.9)

2. Secondary Outcome: Mean Number of Injections.
Description: The average number of intravitreal ranibizumab injections in each arm of the study will be recorded.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Monthly Ranibizumab | Treat and Extend Ranibizumab
Number analyzed (Participants) | 10 | 10
injections | 19.4 (5.9) | 18.8 (2.9)

3. Secondary Outcome: Mean Change in Spectral Domain Optical Coherence Tomography (SD-OCT) Central Foveal Thickness (CFT).
Description: Evaluate the average change in the swelling from diabetic macular edema measured with the optical coherence tomography machine.
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Monthly Ranibizumab | Treat and Extend Ranibizumab
Number analyzed (Participants) | 10 | 10
microns | -169.0 (98.5) | -146.8 (122.0)

4. Secondary Outcome: Percentage of Patients With Best Corrected Visual Acuity (BCVA) Snellen-equivalent of 20/40 or Better.
Description: The percentage of patients with 20/40 vision as assessed by the number of letters read correctly on the ETDRS eye chart at a starting test distance of 20 feet.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Ranibizumab | Treat and Extend Ranibizumab
Number analyzed (Participants) | 10 | 10
Participants | 10 | 9

5. Secondary Outcome: Percentage of Patients Anatomically "Dry."
Description: Spectral domain OCT will be used to check the patients' central foveal thickness at each visit and the percentage with "dry" maculas at months 3,6, and 12 based on spectral domain OCT measurements per the study protocol will be recorded.
Time Frame: 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Monthly Ranibizumab | Treat and Extend Ranibizumab
Number analyzed (Participants) | 10 | 10
Participants | 8 | 7

ADVERSE EVENTS:
Arm/Group | Monthly Ranibizumab | Treat and Extend Ranibizumab
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10 | 1/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monthly Ranibizumab (N=10) | Treat and Extend Ranibizumab (N=10)
Death (Cardiac disorders) | 1 (1) | 0 (0) — Suspected MI
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monthly Ranibizumab (N=10) | Treat and Extend Ranibizumab (N=10)
Vitreous Hemorrhage (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size, single-center, unmasked trial. This pilot study should be interpreted in the context of these limitations, yet may yield some guidance on one of the more common dosing methods for anti-VEGF medications in DME.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes